CLINICAL TRIAL: NCT01053078
Title: Study of the Effect of Naltrexone on Cerebral Blood Flow and Hypoglycemia in Type 1 Diabetes Mellitus
Brief Title: Naltrexone and Hypoglycemia in Type 1 Diabetes
Acronym: Naltrexone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0903M60907; R01DK062440 (NIH); 7-09-DCS-02 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes; Hypoglycemia Unawareness
Keywords: Type 1 diabetes; Hypoglycemia unawareness; low blood sugar
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Naltrexone (Experimental)
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Naltrexone — 1 month treatment; Naltrexone 25mg once daily for 5 days, then 50 mg once daily for 23 days
  Other Names: ReVia
  Arms: Naltrexone
Other: Placebo — 1 month treatment; placebo tablet once daily for 28 days
  Arms: Placebo

SUMMARY:
Low blood sugar is also called hypoglycemia. Usually, it is mild and can be treated quickly and easily by eating or drinking a small amount of a sugar-rich food. If low blood sugar is left untreated, it can get worse and cause confusion, clumsiness or fainting. Severe hypoglycemia can lead to seizures, coma, and even death.

Some people with diabetes do not have early warning signs of low blood sugar. This condition is called hypoglycemia unawareness. It happens when the body stops reacting to low blood sugar levels and the person does not realize that they need to treat their hypoglycemia. This can lead to more severe and dangerous hypoglycemia.

The purpose of this early study is to see if a drug called naltrexone should be studied more in people with Type I diabetes and hypoglycemia unawareness. This study will show whether naltrexone could reduce hypoglycemia unawareness. The study will also show, by using magnetic resonance imaging (also called MRI), whether naltrexone changes the way blood flows in the brain when a person is experiencing hypoglycemia.

DETAILED DESCRIPTION:
Visit 1

This visit is estimated to last approximately 1 hour.

At this visit, you will be asked to complete a questionnaire about hypoglycemia unawareness. Some questions about your medical history may be asked in order to make sure you are eligible to be in this study. You will also have some blood collected for tests that measure how your liver and kidneys are working. A blood test that measures muscle breakdown will also be done. If you are a female who could become pregnant, a pregnancy test will also be done. The amount of blood that will be collected at this visit is approximately three teaspoons. This visit is estimated to last approximately one hour.

You will be asked to wear a continuous glucose monitor (CGMS) around the clock for the seven days before the MRI study. This involves putting a small plastic sensor under the skin on your stomach and carrying the monitor that attaches to the sensor. The sensor measures your glucose and records the readings automatically on the monitor. The monitor is about the size of the palm of a woman's hand. The information stored on the monitor can be sent to a computer that the researcher uses. The researcher will insert the CGMS at visit 1.

Between Visit 1 and Visit 2

You will also be asked to keep careful records for the study every day for the next seven days. You will be asked to check your blood glucose before each of three meals and before you go to sleep at night. You will also be asked to write down your blood glucose levels and bring those records back for the researcher.

Visit 2

Seven days after visit 1 you will be asked to report to the Center for Magnetic Resonance Research (CMRR) at 7:30AM for your first MRI scan. The study will be done in the morning after an overnight fast. All subjects will be asked to fast for a minimum of 8 hours before arriving at the center. The researcher will advise you on how to adjust your insulin regimen during the 1-2 days before the MRI scan to be sure your blood sugar is in good control when you arrive at the CMRR.

Alternatively, you may be asked to come to the Clinical Research Unit the night before the MRI study You will be admitted to the Clinical Research Unit, and stay overnight there. You will not be given any food after your evening meal until your test is completed at about lunch time on the following day. Your evening dose of long-acting insulin or your pump will be held after 6:00 p.m. that evening. Your blood glucose will be measured every 1-2 hours. An intravenous (IV) catheter will be placed in your arm and will stay there until your test is over the next day. You will be given insulin and glucose as needed to keep your blood sugars between 100 and 150 mg/dl through the night leading to testing on the next day. In the morning, you will be transferred to the Center for Magnetic Resonance Research (CMRR) for an MRI.

At the CMRR, an IV will be placed in each of your arms. This will allow for giving insulin, glucose and potassium during the test. A third IV will be placed in one of your legs. This catheter will be put in so that blood can be collected during the test. After the catheter in your leg is placed you will rest for 30 minutes. After thirty minutes, blood will be collected from the catheter in your leg for laboratory tests. The test is then ready to begin.

You will be given insulin through the catheter in one arm and you will be placed in the MRI machine. Your glucose will be checked every five minutes throughout the study. Blood will also be collected every 30 minutes for other laboratory tests. When your glucose drops to 50 mg/dl it will be held at that level for approximately 30 minutes so the measures of blood flow and glucose concentrations in your brain can be taken. While your blood sugar is dropping, you will be asked about any symptoms you may feel. After the measures have been taken, the insulin given through the IV will be stopped and you will be given glucose to bring it back to a normal level.

You will be at the CMRR for 4-6 hours. After the test is completed, your IVs will be taken out, you will resume your usual diabetes treatments, and you will be fed a meal.

Between the time you are admitted to the Clinical Research Unit and the time you are discharged after your MRI test, just less than one cup of blood will be collected.

You will be given a supply of naltrexone, the study medication, or placebo, with instructions for taking the medication over the next four weeks. You will be randomly assigned (like a flip of a coin) to naltrexone, or to a placebo (a pill that does not contain any medicine). Neither you nor your study doctor will know which study treatment (placebo or naltrexone) you are receiving. If it becomes necessary to know for medical reasons, the information will be made available.

Between Visits 2 and 3

While you are taking naltrexone or placebo you will be asked not to use Tylenol (or any other product containing acetaminophen), Advil (or any other product containing ibuprofen or a non-steroidal anti-inflammatory drug), or aspirin. You will also be asked to avoid alcohol while taking naltrexone. If you have any concerns or questions about using these substances during the time you are taking naltrexone please ask the study doctor or coordinator.

You should always take your naltrexone dose right after you eat a meal.

Days 1 - 5: Starting the day after your MRI test, you will be asked to take one 25 mg tablet of naltrexone or placebo each day for the next five days.

Days 6 - 10: On these days you will be asked to take one 50 mg tablet of naltrexone or placebo each day.

Days 11- 14: On these days you will be asked to take one 50 mg tablet of naltrexone or placebo twice each day. Visit 2 for the study will occur on Day 14.

Visit 3

This visit is estimated to last approximately 30 minutes.

You will come to the Clinical Research Unit for a short visit on this day. Blood will be collected for tests that measure how your liver and kidneys are working. A blood test that measures muscle breakdown will also be done. Just like at visit 1, the amount of blood collected from you at this visit will be approximately three teaspoons.

The study doctor or coordinator will also talk to you about how you are feeling. You will be asked about whether you have been taking naltrexone or placebo according to the study plan.

Between Visits 3 and 4

Days 15 - 21: On these days you will be asked to take one 50 mg tablet of naltrexone or placebo twice each day.

Visit 4

This visit is estimated to last approximately 30 minutes.

You will be asked to wear a continuous glucose monitor (CGMS) around the clock for the seven days before the MRI study. This involves putting a small plastic sensor under the skin on your stomach and carrying the monitor that attaches to the sensor. The sensor measures your glucose and records the readings automatically on the monitor. The monitor is about the size of the palm of a woman's hand. The information stored on the monitor can be sent to a computer that the researcher uses. The researcher will insert the CGMS at visit 4.

Between Visits 4 and 5

Days 22 - 28: On these days you will be asked to take one 50 mg tablet of naltrexone or placebo twice each day. You will take your last study dose of naltrexone or placebo on Day 28.

Starting on Day 22, just like in the first part of this study, you will also be asked to keep careful records for the study every day during this time. You will be asked to check your blood glucose before each of three meals and before you go to sleep at night. You will also be asked to write down your blood glucose levels and bring those records back for the researcher.

Visit 5

Just like in the first part of the study, you will be asked to report to the Center for Magnetic Resonance Research (CMRR) at 7:30AM for your first MRI scan. The study will be done in the morning after an overnight fast. All subjects will be asked to fast for a minimum of 8 hours before arriving at the center. The researcher will advise you on how to adjust your insulin regimen during the 1-2 days before the MRI scan to be sure your blood sugar is in good control when you arrive at the CMRR.

Alternatively, you will be asked to come to the Clinical Research Unit the night before the MRI study. You will come in the day before you take your last dose of naltrexone or placebo. You will be admitted to the Clinical Research Unit, and stay overnight there. You will not be given any food after your evening meal until your test is completed at about lunch time on the following day. Your evening dose of long-acting insulin or your pump will be held after 6:00 p.m. that evening. Your blood glucose will be measured every 1-2 hours. An intravenous (IV) catheter will be placed in your arm and will stay there until your test is over the next day. You will be given insulin and glucose as needed to keep your blood sugars between 100 and 150 mg/dl through the night leading to testing on the next day. In the morning, you will be transferred to the Center for Magnetic Resonance Research (CMRR) for an MRI.

Blood will be collected for tests that measure how your liver and kidneys are working. A blood test that measures muscle breakdown will also be done.

The procedures for Visit 5 will be exactly the same as the procedures in Visit 2. The only difference is that you will not be given any naltrexone or placebo at the end of the visit. When you complete Visit 5, your participation in the study has been completed.

At the CMRR, an IV will be placed in each of your arms. This will allow for giving insulin, glucose and potassium during the test. A third IV will be placed in one of your legs. This catheter will be put in so that blood can be collected during the test. After the catheter in your leg is placed you will rest for 30 minutes. After thirty minutes, blood will be collected from the catheter in your leg for laboratory tests. The test is then ready to begin.

You will be given insulin through the catheter in one arm and you will be placed in the MRI machine. Your glucose will be checked every five minutes throughout the study. Blood will also be collected every 30 minutes for other laboratory tests. When your glucose drops to 50 mg/dl it will be held at that level for approximately 30 minutes so the measures of blood flow and glucose concentrations in your brain can be taken. While your blood sugar is dropping, you will be asked about any symptoms you may feel. After the measures have been taken, the insulin given through the IV will be stopped and you will be given glucose to bring it back to a normal level.

You will be at the CMRR for 4-6 hours. After the test is completed, your IVs will be taken out, you will resume your usual diabetes treatments, and you will be fed a meal.

Between the time you are admitted to the Clinical Research Unit and the time you are discharged after your MRI test, just less than one cup of blood will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Type 1 diabetes
* Hypoglycemia unawareness
* Capable of providing informed consent

Exclusion Criteria:

* Concomitant regular use of acetaminophen, aspirin or ibuprofen
* History of drug or alcohol abuse
* Psychiatric illness
* Elevations in ALT (Alanine Aminotransferase), AST (Aspartate Aminotransferase), creatinine or history of hepatitis, liver failure, or renal failure/insufficiency
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Seaquist, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Olawsky E, Zhang Y, Eberly LE, Helgeson ES, Chow LS. A New Analysis Tool for Continuous Glucose Monitor Data. J Diabetes Sci Technol. 2022 Nov;16(6):1496-1504. doi: 10.1177/19322968211028909. Epub 2021 Jul 20. PMID 34282646
- [Derived] Moheet A, Mangia S, Kumar A, Tesfaye N, Eberly LE, Bai Y, Kubisiak K, Seaquist ER. Naltrexone for treatment of impaired awareness of hypoglycemia in type 1 diabetes: A randomized clinical trial. J Diabetes Complications. 2015 Nov-Dec;29(8):1277-82. doi: 10.1016/j.jdiacomp.2015.08.004. Epub 2015 Aug 12. PMID 26345338

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 14 | 15
Completed | 10 | 12
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (13) | 39 (10) | 42 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Blood Flow
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: percentage of signal intensity change
Groups:
- Naltrexone: Double blind placebo comparable
  Naltrexone: 1 month treatment
  Naltrexone: Naltrexone 25 mg once daily with dose escalation to 50 mg BID to day 28
- Placebo: Naltrexone: 1 month treatment
  Naltrexone: Naltrexone 25 mg once daily with dose escalation to 50 mg BID to day 28
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 10 | 12
percentage of signal intensity change | 1.7 (1.9) | 1.3 (3.3)

2. Secondary Outcome: Hypoglycemia Symptom Score
Description: Hypoglycemia symptom score is determined by a standardized 12-item questionnaire. Participants rank hypoglycemic symptoms on a Likert scale from 0 (no symptoms) to 6 (severe symptoms). Total score is a sum of the 12 items scores with a total score range from 0 to 72. Higher scores indicated increased severity of symptoms associated with hypoglycemia.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 10 | 12
score on a scale | 12.6 (7.5) | 14.5 (12.2)

ADVERSE EVENTS:
Arm/Group | Naltrexone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 3/10 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone (N=10) | Placebo (N=12)
headache (Nervous system disorders) | 3 | 0
diarrhea (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT01053078/Prot_SAP_000.pdf